CLINICAL TRIAL: NCT05792176
Title: A Randomized Controlled Trial of Ukulele Playing Compared to Music Listening to Improve Cognition in People with Multiple Sclerosis: a Feasibility Study
Brief Title: Ukulele Playing to Improve Cognition in People with Multiple Sclerosis: a Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Carolyn Phillips, Assistant Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STUDY00003870
Record Dates: First submitted 2023-02-16; First posted 2023-03-31 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-11

CONDITIONS: Multiple Sclerosis; Pathologic Processes; Demyelinating Autoimmune Diseases, CNS; Autoimmune Diseases of the Nervous System; Nervous System Diseases; Demyelinating Diseases; Autoimmune Diseases; Immune System Diseases
Keywords: cognitive rehabilitation
MeSH Terms: conditions — Multiple Sclerosis; Pathologic Processes; Demyelinating Autoimmune Diseases, CNS; Autoimmune Diseases of the Nervous System; Nervous System Diseases; Demyelinating Diseases; Autoimmune Diseases; Immune System Diseases

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Musical Training Intervention (Experimental): Participants randomized to this arm receive a 12-week intervention to teach them how to play the ukulele. The ukulele is a very manageable instrument to learn and requires less hand dexterity than other stringed instruments. Each week participants will follow the musical training intervention (MTI) protocol that provides instruction on how to tune, hold, and strum the ukulele and play basic chords. To practice the chords, they will also learn popular songs (e.g., Chain of Fools, Three Little Birds, Happy Birthday, Don't Worry Be Happy, and Stand by Me). Participants will be instructed to follow each session outlined weekly and asked to practice the instrument for at least 30 minutes, 5 days a week. They will be given a paper and digital version of the MTI protocol. A member of our research team will call the participants weekly to answer any questions about the MTI protocol.
  Interventions: Behavioral: Music Training Intervention
- Music Listening (Active Comparator): Participants randomized to this arm will be asked to listen to their preferred music for at least 30 minutes, 5 days a week. A member of our research team will call them every week to answer any questions they have about the ML protocol. They will be asked to record their experience in a practice log.
  Interventions: Behavioral: Music Listening

INTERVENTIONS:
Behavioral: Music Training Intervention — The Music Training Intervention (MTI) entails 12-weeks of online instruction to learn to play the ukulele. Participants will be taught the basic information on how to handle and hold the ukulele, musical chords, and popular songs. They will be instructed to play at least 30-minutes a day, five days a week.
  Arms: Musical Training Intervention
Behavioral: Music Listening — Participants randomized to this arm will be asked to listen to their preferred music for at least 30 minutes, 5 days a week. A member of our research team will call them every week to answer any questions they have about the ML protocol. They will be asked to record their experience in a practice log.
  Arms: Music Listening

SUMMARY:
Over the past 10 years, the rates of multiple sclerosis (MS) have nearly doubled in the United States. This chronic, neuroinflammatory, and neurodegenerative disease is most often diagnosed between the ages of 20-40. Cognitive impairment effects up to 70% of people with MS (PwMS) and has a detrimental impact on mental health, social connections, and employment. Further, up to 50% of PwMS also struggle with depression. Numerous cognitive rehabilitation programs are available to address cognitive impairment, but few interventions have simultaneous effects on cognition and emotional well-being. Music interventions have potential to fill this gap. Brain imaging studies on music and emotion show that music can modulate activity in the brains structures that are known to be crucially involved in emotion. Further, music engages areas of the brain that are involved with paying attention, making predictions, and updating events in our memory.

The purpose of this study is to determine the feasibility of an online musical training intervention (MTI) for PwMS and explore the potential effect on cognition, psychosocial, and functional well-being compared to an active control group (music listening (ML)). The specific aims are to: 1) determine the feasibility and acceptability of delivering the MTI virtually over three months to PwMS; 2) evaluate the effect of the MTI on cognitive functioning (processing speed, working memory, cognitive flexibility, response inhibition), psychosocial (anxiety, depression, stress, quality of life, self-efficacy) and functional (insomnia) well-being compared to ML; and 3) (exploratory aim) to utilize non-invasive neuroimaging to determine if pre-intervention brain activity predicts post-intervention cognitive functioning.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) affects more than 2.8 million people worldwide. The prevalence has increased in every region worldwide since 2013, and in the United States, rates have nearly doubled. It is the main cause of nontraumatic disability in young adults in many countries. MS is a chronic neuroinflammatory and neurodegenerative disease with an unpredictable course. Varying visible and invisible symptoms occur in MS. The invisible symptoms, such as fatigue, depression, psychological distress, insomnia, and cognitive dysfunction pose a significant burden on quality of life (QoL) and workforce participation, rendering PwMS more vulnerable to mental health challenges compared to those affected by physical disability alone. Cognitive impairment occurs in 40-70%, depression in up to 50%, and fatigue can be present in up to 85-95% of PwMS. The interplay of cognitive impairment, mood, impaired sleep quality, and fatigue contributes significantly to worsened QoL. Cognitive impairment can occur in early and late phases of the disease and may include alterations in information processing, attention, executive functions and working memory. Multiple interventions have been created to address cognitive impairments such as conventional cognitive rehabilitation, computer-based programs, non-invasive brain stimulation, and neurologic music therapy. Many of these interventions have shown improvements in various domains of cognitive impairment. However, the effect of cognitive rehabilitation on psychosocial well-being in addition to cognitive symptoms is rare.

This research aims to fill a gap in cognitive rehabilitation with an innovative music training intervention for PwMS. Active music engagement interventions (i.e., instrument playing) have shown improvements in cognitive, motor, and psychosocial outcomes in other neurological conditions. However, few studies have examined the impact for PwMS. Most music intervention studies in PwMS evaluate the impact of music on fatigue, pain, mood disorders, walking, and balance. The impact of music on cognition is much less studied. Our team is currently conducting a systematic review examining the differences between active and passive music engagement in PwMS. Sixteen studies were included in the review. Only two studies examined active music making (singing or musical instrument playing), only one of those evaluated the impact on cognition (no improvement), and neither evaluated the effect on psychosocial (anxiety, depression, quality of life) outcomes. Twelve of the studies evaluated passive music engagement (music listening with or without movement); however, the primary outcome in most of these studies was neurological motor skills versus non-motor or psychosocial outcomes. One study, that used both active and passive musical engagement, examined the effect of cognitive rehabilitation plus neurological music therapy on cognitive abilities, mood, emotional components, and MS quality of life. They found significant improvements in cognitive function, motivation, emotional awareness, depression, and quality of life in the intervention that entailed cognitive rehabilitation plus neurological music therapy. However, no significant differences were found between the experimental group (cognitive rehabilitation plus neurological music therapy) and active control (cognitive rehabilitation alone).

Music listening and making is processed throughout spinal, subcortical, and cortical regions, and thus has meaningful and broad impacts on complex cognitive, affective, and sensorimotor processes. The impact of instrumental music playing on executive functioning has been demonstrated in many studies with children; however, this has not been studied in PwMS. Specific to executive function, neuroimaging studies with functional magnetic resonance imaging (fMRI) and functional near-infrared spectroscopy (fNIRS) show an increase in neural activations the right frontal and prefrontal regions in PwMS on cognitive tests requiring lower cognitive load (e.g., 1-back) working memory tasks when compared to healthy controls and lower activation on higher cognitive load tasks (2- and 3-back). Theoretically, it is hypothesized that the neuronal damage caused by MS causes processing resources to be diminished, thus different brain areas are recruited to cope with task demands as difficulty increases. The rehabilitative effects of music in relation to other neurological disorders is linked to changes in brain neuroplasticity, which describes the adaption and cortical reorganization after training or learning a new task. This study will examine the feasibility of an online musical training intervention (MTI) for PwMS, explore the potential effect on cognitive functioning, psychosocial, and functional well-being, and explore a neuroimaging via fNIRS, a non-invasive technique, to determine if pre-intervention brain activity predicts post-intervention cognitive functioning.

The purpose of this study is to determine the feasibility of an online musical training intervention (MTI) for PwMS and explore the potential effect on cognition, psychosocial, and functional well-being compared to an active control group (music listening (ML)). The specific aims are to: 1) determine the feasibility and acceptability of delivering the MTI virtually over three months to PwMS; 2) evaluate the effect of the MTI on cognitive functioning (processing speed, working memory, cognitive flexibility, response inhibition), psychosocial (anxiety, depression, stress, quality of life, self-efficacy) and functional (insomnia) well-being compared to ML; and 3) (exploratory aim) to utilize non-invasive neuroimaging to determine if pre-intervention brain activity predicts post-intervention cognitive functioning.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with multiple sclerosis (relapsing remitting, secondary progression, primary progressive)
* Diagnosed more than 6 months prior to starting study
* Self-reported cognitive impairment as assessed by having at least 5 problems "sometimes" or more often on the Perceived Deficits Questionnaire
* Read, write, and understand English
* Access to computer and zoom

Exclusion Criteria:

* Diagnosed with another neurological condition that causes cognitive impairment
* MS exacerbation within the last 30 days
* Unable to travel to The University of Texas at Austin for fNIRS data collection
* Professional musician (primary source of income)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Intervention Feasibility | Immediately post-intervention
  Feasibility will be evaluated by tracking the percentage of participants screened and enrolled.
Intervention Feasibility | Immediately post-intervention
  Feasibility will be evaluated by tracking the average number of participants enrolled monthly.
Intervention Feasibility | Immediately post-intervention
  Protocol adherence will be evaluated by recording the average number of modules completed by participants.
Intervention Acceptability | Immediately post-intervention
  Acceptability will be evaluated with semi-structured interview questions to understand the participant's perception of MTI delivery and content and the perceived impact.

SECONDARY OUTCOMES:
Mean Change from Baseline in Anxiety Scores at 12 weeks and 16 weeks | Immediately post-intervention and 1-month post-intervention
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Distress-Anxiety Short-Form 8a will be used. The minimum score is 8, and the maximum score is 40. Higher scores indicate more anxiety.
Mean Change from Baseline in Depression Scores at 12 weeks and 16 weeks | Immediately post-intervention and 1-month post-intervention
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Short-Form 8a will be used. The minimum score is 8, and the maximum score is 40. Higher scores indicate higher levels of depressive symptoms.
Mean Change from Baseline in Stress Scores at 12 weeks and 16 weeks | Immediately post-intervention and 1-month post-intervention
  The Perceived Stress Scale will be used. The minimum score is 0, and the maximum score is 40. Higher scores indicate more perceived stress.
Mean Change from Baseline in Self-Efficacy Scores at 12 weeks and 16 weeks | Immediately post-intervention and 1-month post-intervention
  The Chronic Disease Self-Efficacy Scale will be used. The minimum score is 6, and the maximum score is 60. Higher scores indicate more self-efficacy.
Mean Change from Baseline in Quality of Life Scores at 12 weeks and 16 weeks | Immediately post-intervention and 1-month post-intervention
  The Multiple Sclerosis Quality of Life Questionnaire will be used. The minimum score is 27, and the maximum score is 135. Higher scores indicate worse quality of life.
Mean Change from Baseline in Sleep Disturbance Scores at 12 weeks and 16 weeks | Immediately post-intervention and 1-month post-intervention
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep disturbance Short-Form 6a will be used. The minimum score is 6, and the maximum score is 30. Higher scores indicate more sleep disturbance.
Mean Change from Baseline in Attention Scores at 12 weeks and 16 weeks | Immediately post-intervention and 1-month post-intervention
  The Trail Making A&B will be used to measure attention. Trails A and B are two separate timed tests. Faster time means greater attention.
Mean Change from Baseline in Memory Scores at 12 weeks and 16 weeks | Immediately post-intervention and 1-month post-intervention
  Immediate and delayed recognition tests will be used. Participant are shown 10 words to memorize. In the immediate recognition test, they are immediately asked to identify the 10 words they memorized out of a list of 20. Later in the testing series, participants will again be asked to recall the 10 words. The number of correct responses will be scored. Higher scores means better memory.
Mean Change from Baseline in Executive Functioning Scores at 12 weeks and 16 weeks | Immediately post-intervention and 1-month post-intervention
  The Digit-Symbol Substitution will be used to measure processing speed and accuracy to evaluate executive functioning. In this test, participants match arbitrary symbols to digits. Scores are calculated by the number of trials correctly completed in 60 seconds.
Mean Change from Baseline in Executive Functioning Scores at 12 weeks and 16 weeks | Immediately post-intervention and 1-month post-intervention
  The Stroop Color and Word Test evaluates impulse control and inhibition to evaluate executive functioning. When the name of a color (e.g., "blue," "green," or "red") is displayed in an incongruent color, name (for example, the word "blue" printed in red), naming the color of the word takes longer and is more prone to errors than when the word and color are congruent or neutral. The scoring uses median duration of incongruent trials.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Phillips, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No